CLINICAL TRIAL: NCT03214965
Title: The Use of the Social Networking to Promote Educational and Consultative Actions Among Kidney Transplanted Adolescents. Comparison of the Knowledge, Satisfaction and Self-esteem Between Two Groups: a Randomized Clinical Trial.
Brief Title: The Use of the Social Networking to Promote Educational and Consultative Actions Among Kidney Transplanted Adolescents.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Claudiana Briskiewski Pase, Registered Nurse, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5259/16
Record Dates: First submitted 2016-09-19; First posted 2017-07-12 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Kidney Transplantation; Education
Keywords: Kidney transplantation; Facebook; Education; Adolescent; Social Networking

STUDY DESIGN:
Intervention Model Description: Participants are assigned to participate into one of two groups (control group or intervention group) in parallel for the duration of the study. The control group receives no form of intervention or education. The intervention group participates into a closed facebook group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facebook group (Active Comparator): Patients of the kidney transplantation group randomly assigned to be part of a closed facebook group.
  Interventions: Behavioral: Facebook group
- Control group (No Intervention): Patients of the kidney transplantation group that do not receive specific educational interventions.

INTERVENTIONS:
Behavioral: Facebook group — A closed facebook group used to deliver multimedia content specifically produced to inform the participants about chronic kidney disease, kidney transplantation and related topics. This group is also used to share doubts and life experiences among participants and the interdisciplinary team.
  Arms: Facebook group

SUMMARY:
This study is designed to compare the knowledge, satisfaction and self-esteem of kidney transplanted adolescents measured through questionnaires between two groups: patients undergoing conventional treatment with no other intervention versus patients undergoing conventional treatment and receiving additional educational and consultative actions using a closed facebook group.

DETAILED DESCRIPTION:
Based on literature, there are strong evidences that the use of social media improves the outcomes of chronic treatments. Currently, there is no study using social media as an education tool in kidney transplant patients in Brazil. This study is designed to answer the question: "Does the use of a popular social media such as facebook improves the knowledge, satisfaction and self-steem levels among kidney transplant adolescents when compared with their peers ?" This is a non-blinded randomized clinical trial. Patients will be randomly included into one of the two groups: the control group who will not receive any intervention or the facebook group (who will receive additional educational and consultative support through a closed facebook group) After three months, knowledge level, satisfaction level and self-esteem will be assessed by specific designed questionnaires and by the application of the Rosenberg's self-esteem scale. The study will have a sample of 122 subjects, equally divided (61 participants in each group). Collected data will be compared using the chi square test.

ELIGIBILITY:
Inclusion criteria

* patients receiving follow up care by the transplant interdisciplinary team either in the pre or in the post transplant period

Exclusion criteria

* patients with chronic kidney disease not enrolled to receive a kidney transplant.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Knowledge about the disease | 3 months
  Knowledge about the disease and associated conditions measured by a specific designed questionnaire.
Satisfaction about the treatment | 3 months
  Satisfaction with the interdisciplinary team obtained by a specific designed questionnaire
Self-esteem | 3 months
  Assessment of the participant's self-esteem through the application of the "Rosenberg's Self-Esteem Scale"

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Goldmeier, PhD, Study Director — Fundação Instituto de Cardiologia
Locations (1):
- Hospital da Criança Santo Antônio da Santa Casa de Misericórdia, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared among other researchers.

REFERENCES:
- [Background] Sesso, R. Epdemiologia da doença renal crônica no Brasil. Guia de Nefrologia. São Paulo: Manole; 2002.
- [Background] Garcia, VD, Pacheco, L. Revista Brasileira de transplantes: Dimensionamento dos transplantes no Brasil e em cada estado. Ano XX n. 4. 2014.
- [Background] Lira ALBC, Guedes MVC, Lopes MVO. Adaptação psicossocial do adolescente pós-transplante renal segundo a teoria de roy. Invest Educ Enferm. 2005; 23;1: 68-77.
- [Background] Morales LC, Castilho E. Vivencias de los(as) adolescentes en diálisis: una vida con múltiples pérdidas pero con esperanza. Colombia Médica. 2007; 38; 4: 44-53.
- [Background] Pereira L M. Adesão ao tratamento imunossupressor no transplante renal. São Paulo: Permanyer Brasil Publicações, Ltda; 2012.
- [Background] Garcez JLAF, Maciel FR, Cardoso VMB. Considerações ergonômicas para aplicação de mídia em ambientes educacionais para crianças de ensino fundamental. Produção. 2012; 22; 2: 284-295.
- [Background] Vitola, SP. Transplante renal em crianças com peso inferior a 15 Kg; acesso cirúrgico extraperitoneal- Experiência em 62 transplantes. [Tese]. Porto Alegre: Pós-graduação em Ciências Cirúgicas da Faculdade de Medicina da Universidade Federal do Rio Grande do Sul, 2011.
- [Background] Casas RV. Transplante renal pediátrico. Enero, 2003; 59; 1460, 24-30.
- [Background] Garcia CD, Bittencourt VB, Rohde RW, Vitola SP. Transplante renal pediátrico. in: Garcia CD, Pereira JD, Zago MK, Garcia VD. Manual de doação e transplantes. 1.ed. Rio de Janeiro: Elsevier; 2013. p. 225-234.
- [Background] Goldani JC, Vitola SP, Souza LV, Souza LVB. Transplante renal. In: Garcia CD, Pereira JD, Zago MK, Garcia VD. Manual de doação e transplantes. 1.ed, Rio de Janeiro: Elsevier; 2013. p. 193-198.
- [Background] Matas AJ. Impacto de não-adesão do receptor nos desfechos em longo prazo de transplante. Revisão da literatura e experiência da universidade de Minnesola. Bras. Transpl. 2007; 828-831.
- [Background] Nifa S, Rudnicki T. Depressão em pacientes Renais Crônicos em tratamento de Hemodiálise. Rev SBPH. 2010; 13; 1.
- [Background] Brasil, Secretaria da Saúde. Manual de atenção à saúde do adolescente/ Secretaria da Saúde. Coordenação de Desenvolvimento de Programas e Políticas de Saúde- CODEPPS. São Paulo: SMS, 2006. 328p
- [Background] Marciano RC. Transtornos mentais e qualidade de vida em crianças e adolescentes com doença renal crônica em seus cuidadores.[dissertação]. Minas Gerais: Pós-graduação da Faculdade de Medicina da UFMG, 2009.
- [Background] Christensen CM. Inovação na gestão da saúde: soluções disruptivas para reduzir custos e aumentar qualidade. Porto Alegre: Bookman, 2009. 422p.
- [Background] Stoltz T. Mídia, cognição e educação. Educar. 2005; 26; 147-156.
- [Background] Garcez JLAF, Maciel FR, Cardoso VMB. Considerções ergonômicas para aplicação de mídia em ambientes educacionais para crianças de ensino fundamental. Produção. 2012; 22; 2. 284-295.
- [Background] Lenhart A. Teens and Mobile Phones. Pew Internet & American Life Project. 2010.
- [Background] Nielsen. Social media comes of age. Retrieved May 2 2013 from <http://www.nielsen.com/us/en/newswire/2012/social-media-report-2012-social-media-comes-of-age.html>.
- [Background] Barbosa SM, Dias FLA, Pinheiro AKB, Pinheiro PNC, Vieira NFC. Jogo educativo como estratégia de educação em saúde para adolescentes na prevenção às DST/AIDS. Rev. Eletr. Enf. 2010; 12; 2. 337-41.
- [Background] Ellison N, Steinfield C, Lampe C. The Benefits of Facebook ''Friends:'' Social Capital and College Students' Use of Online Social Network Sites. Journal of Computer-Mediated Communication. 2007; 12. 1143-1168.
- [Background] Brasil. Ministério da Saúde. Conselho Nacional de Saúde. Resolução 196/96, de 10 de Outubro de 1996. Dispõe sobre as diretrizes e normas regulamentadoras de pesquisa envolvendo seres humanos. Brasília, 1996.
- [Background] Gamonar F. A morte dos Shoppings, o fim do fecebook e o futuro criado pelos millennials. 2015. https://www.linkedin.com/pulse/morte-dos-shoppings-o-fim-do-facebook-e-futuro-criado-flavia-gamonar. Visualizado dia: 14/02/16.
- [Background] Carmo EH, Barreto ML, Silva JBJ. Mudanças nos padrões de morbimortalidade da populaçãoo brasileira: os desafios para um novo século. Epidemiol. Serv. Saúde. 2003; 12. 2. 63-75.
- [Background] Randomization.com [internet]. Available in:http:// www.randomization.com
- [Background] Dini GM, Quaresma MR, Ferreira LM. Adaptação cultural e validaçãoo da versão Brasileira da Escala de Auto-estima de Rosenberg.Rev. Soc. Bras. Cir. Plast. 2004; 19. 1. 41-52.
- [Background] Rosenberg M. Society and the adolescente self image. Princeton: Princeton university Press; 1965.
- [Background] Noronha IL, Ferraz AS, Silva AP Filho, Saitovich D, Carvalho DBM, Paula FJ, Campos H, Lanhez LE, Garcia VD. Transplante Renal: Doador e Receptor. Projeto Diretrizes Associação Médica Brasileira e Conselho Federal de Medicina. 1-19.
- [Result] Oliva M, Singh TP, Gauvreau K, Vanderpluym CJ, Bastardi HJ, Almond CS. Impact of medication non-adherence on survival after pediatric heart transplantation in the U.S.A. J Heart Lung Transplant. 2013 Sep;32(9):881-8. doi: 10.1016/j.healun.2013.03.008. Epub 2013 Jun 4. PMID 23755899
- [Result] Takemoto SK, Pinsky BW, Schnitzler MA, Lentine KL, Willoughby LM, Burroughs TE, Bunnapradist S. A retrospective analysis of immunosuppression compliance, dose reduction and discontinuation in kidney transplant recipients. Am J Transplant. 2007 Dec;7(12):2704-11. doi: 10.1111/j.1600-6143.2007.01966.x. Epub 2007 Sep 14. PMID 17868065
- [Derived] Pase C, Mathias AD, Garcia CD, Garcia Rodrigues C. Using Social Media for the Promotion of Education and Consultation in Adolescents Who Have Undergone Kidney Transplant: Protocol for a Randomized Control Trial. JMIR Res Protoc. 2018 Jan 9;7(1):e3. doi: 10.2196/resprot.8065. PMID 29317381